CLINICAL TRIAL: NCT04173351
Title: The Effects of Antenatal Education and Counseling on Childbirth Fear of Nulliparous Women and Their Attitudes Towards Childbirth
Brief Title: The Effects of Antenatal Education and Counseling on Childbirth Fear of Nulliparous Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 50687469-1491
Record Dates: First submitted 2019-11-20; First posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Fear of Childbirth
Keywords: childbirth; nulliparous; childbirth fear; antenatal education; counseling; attitude; pain
MeSH Terms: conditions — Behavior; Pain | interventions — Educational Status; Counseling

STUDY DESIGN:
Intervention Model Description: This randomized controlled study was conducted at Gulhane Training and Research Hospital, Obstetrics and Gynecology clinic between February 2016 and January 2017. The CONSORT (Consolidated Standards of Reporting Trials) guidelines for reporting randomised controlled trials (RCTs) has been used to describe the methods.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pregnant women in intervention group completed the PIQ, W-DEQ-A and CAQ between the 28th and the 34th gestational weeks. Date of the next antenatal follow-up of the participants in the intervention group was recorded and they were given an appointment for the antenatal education. Women, whose date of next antenatal follow-up was unknown, were asked to inform the researchers about their appointment. Following the antenatal follow-up, the pregnant women in the intervention group were given an antenatal childbirth education and an educational brochure after the education. Also, provided telephone counseling to the intervention group one week after the education. Participants in the intervention group filled the W-DEQ-A and CAQ during the 38th and the 40th gestational weeks. Finally, were completed the W-DEQ-B during the first and the second postnatal days.
  Interventions: Behavioral: Education and Counseling
- Control (No Intervention): Pregnant women in control group completed the PIQ, W-DEQ-A and CAQ between the 28th and the 34th gestational weeks. Participants in the control group filled the W-DEQ-A and CAQ during the 38th and the 40th gestational weeks. Finally, were completed the W-DEQ-B during the first and the second postnatal days.

INTERVENTIONS:
Behavioral: Education and Counseling — Following the pretests between the 28th and the 34th gestational weeks, nulliparous women in the intervention group received a presentation on childbirth preparation at a room of the obstetrics clinic. The education was completed in two sections in a single day. Each session took about 45 minutes there was a 15-minute break between the sessions. Following the education, the questions of the participants were responded and educational brochures on childbirth preparation were given to the participants. One of the researchers of this study telephoned the participant women in the intervention group one week after the childbirth education and provided counseling service about the demands and the points that the nulliparous women wondered.
  Arms: Intervention

SUMMARY:
This study investigates the effects of antenatal education and counseling on childbirth preparation and pain management given to nulliparous women during the last trimester on their childbirth fear and childbirth attitudes.

DETAILED DESCRIPTION:
Pregnancy is an important period of life that the pregnant women have biological, physiological, emotional and social changes in order to adapt to maternity. Fear of childbirth is a common problem and has a negative impact on the childbirth experience. The prevalence of fear associated with childbirth is around 20% but approximately 6 to 10% of women experience intense fear of labour. In Turkey, it estimated that the prevalence of childbirth fear among the Turkish pregnant women was approximately 21% . Fear of childbirth can cause significant problems during childbirth and the postpartum period. This fear is commonly associated with concern for the baby, pain in childbirth, longer first and second stage of labour and dissatisfaction with the childbirth experiences. Especially nulliparous women experience fear of childbirth more than multipar women. Fear of childbirth has also been implicated in women's requests for caesarean sections and increased rate of elective caesarean sections. Antenatal education is an essential health service throughout the world. Antenatal education during the last trimester may decrease childbirth fear. Also, pregnant women who received antenatal education, had a positive birth experience, better maternal adjustment and fewer symptoms of postnatal depression. The aim of this study was to investigate the effects of antenatal education and counseling on childbirth preparation and pain management given to nulliparous women during the last trimester on their childbirth fear and childbirth attitudes.

This randomized controlled study was conducted at Gulhane Training and Research Hospital, Obstetrics and Gynecology clinic between February 2016 and January 2017. 132 nulliparous women between the 28th and 34th gestational weeks constituted the sample of the study. Data was collected by using personal information questionnaire, the Wijma Delivery Expectancy/Experience Questionairre (W-DEQ) Version A, W-DEQ Version B, and Childbirth Attitudes Questionairre (CAQ). Following the pretest, participants in the intervention group received childbirth preparation education and telephone counseling. Participants in the control group received no intervention other than the routine antenatal follow-up. For both groups, pretest and posttest were conducted during the same days, antenatal evaluation took place between the 38th and the 40th gestational weeks and postnatal evaluation was conducted during the first and the second postnatal days. The IBM SPSS (Statistical package for the Social Sciences) 22.0 package program was used to evaluate the data obtained in the study.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparity
* 28-34th gestational age
* Single fetus
* not receive IVF treatment
* Normal vaginal birth

Exclusion Criteria:

* Caesarean section

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Nulliparous pregnant women
Enrollment: 132 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-01-15 (Actual)

PRIMARY OUTCOMES:
Wijma Delivery Expectancy/Experience Questionairre (Version A) (W-DEQ-A) | 10 minutes
  Participants filled before and after education and counseling W-DEQ-A was developed by Klaas and Barbro Wijma in Sweden in 1998. Cronbach's alpha of the scale was 0.88 for primiparous women. The scale consisted of 33 items, which are rated on a six-point Likert type scale (zero=do not agree; five=totally agree). Items 2, 3, 6, 7, 8, 11, 12, 15, 19, 20, 24, 25, 27 and 31 were reverse-scored to calculate the women's individual total score. Higher scores indicated greater fear that the pregnant women experienced. Cutting score of the questionnaire was 85.
Wijma Delivery Expectancy/Experience Questionairre (Version B) (W-DEQ-B) | 10 minutes
  Participants filled on the first and second days of postpartum W-DEQ-B was developed by Klaas and Barbro Wijma in 1998 in order to determine postpartum pains and the feelings and thoughts of women after childbirth. The questionnaire included 32 items rated on a six-point Likert type scale (zero=not at all; five=extremely). Items 2, 3, 6, 7, 10, 11, 14, 18, 19, 23, 24, 26, and, 30 were reverse scored and higher scores indicated greater postnatal fear of childbirth. The questionnaire had six subscales, namely, concerns about labor pain, loneliness, lack of positive feelings, concerns about childbirth, and concerns about baby.
Childbirth Attitudes Questionnaire (CAQ) | 5 minutes
  Participants filled before and after education and counseling CAQ was developed by Lowe in 2000 in order to measure the fear of childbirth. Cronbach's alpha of the scale was 0.83. The questionnaire included 16 items rated on a four-point Likert type scale. Higher scores indicated greater fear.

CONTACTS AND LOCATIONS:
Overall Officials: Gulten Guvenc, Prof. Dr., Principal Investigator — University of Health Sciences, Gulhane Faculty of Nursing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rouhe H, Salmela-Aro K, Toivanen R, Tokola M, Halmesmaki E, Ryding EL, Saisto T. Group psychoeducation with relaxation for severe fear of childbirth improves maternal adjustment and childbirth experience--a randomised controlled trial. J Psychosom Obstet Gynaecol. 2015;36(1):1-9. doi: 10.3109/0167482X.2014.980722. Epub 2014 Nov 24. PMID 25417935
- [Background] Gokce Isbir G, Inci F, Onal H, Yildiz PD. The effects of antenatal education on fear of childbirth, maternal self-efficacy and post-traumatic stress disorder (PTSD) symptoms following childbirth: an experimental study. Appl Nurs Res. 2016 Nov;32:227-232. doi: 10.1016/j.apnr.2016.07.013. Epub 2016 Jul 30. PMID 27969033
- [Background] Hauck YL, Stoll KH, Hall WA, Downie J. Association between childbirth attitudes and fear on birth preferences of a future generation of Australian parents. Women Birth. 2016 Dec;29(6):511-517. doi: 10.1016/j.wombi.2016.05.001. Epub 2016 May 24. PMID 27233945
- [Background] Haapio S, Kaunonen M, Arffman M, Astedt-Kurki P. Effects of extended childbirth education by midwives on the childbirth fear of first-time mothers: an RCT. Scand J Caring Sci. 2017 Jun;31(2):293-301. doi: 10.1111/scs.12346. Epub 2016 Jul 21. PMID 27439382
- [Background] Fenwick J, Toohill J, Gamble J, Creedy DK, Buist A, Turkstra E, Sneddon A, Scuffham PA, Ryding EL. Effects of a midwife psycho-education intervention to reduce childbirth fear on women's birth outcomes and postpartum psychological wellbeing. BMC Pregnancy Childbirth. 2015 Oct 30;15:284. doi: 10.1186/s12884-015-0721-y. PMID 26518597
- [Background] Deliktas A, Kukulu K. Pregnant Women in Turkey Experience Severe Fear of Childbirth: A Systematic Review and Meta-Analysis. J Transcult Nurs. 2019 Sep;30(5):501-511. doi: 10.1177/1043659618823905. Epub 2019 Jan 17. PMID 30651038
- [Background] Karabulut O, Coskuner Potur D, Dogan Merih Y, Cebeci Mutlu S, Demirci N. Does antenatal education reduce fear of childbirth? Int Nurs Rev. 2016 Mar;63(1):60-7. doi: 10.1111/inr.12223. Epub 2015 Nov 27. PMID 26612181
- [Derived] Bektas Pardes B, Guvenc G. The effects of antenatal education and telephone counseling on childbirth fear of nulliparous women and their attitudes toward childbirth: a randomized controlled trial. Rev Assoc Med Bras (1992). 2025 Mar 17;71(1):e20241147. doi: 10.1590/1806-9282.20241147. eCollection 2025. PMID 40105556